CLINICAL TRIAL: NCT04801329
Title: KOREAN POST-MARKETING SURVEILLANCE VYNDAMAX (Registered) CAPSULES FOR THE TREATMENT OF TRANSTHYRETIN AMYLOID CARDIOMYOPATHY (ATTR-CM)
Brief Title: Korean Post-marketing Surveillance Vyndamax® Capsules for the Treatment of Transthyretin Amyloid Cardiomyopathy
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461080; Vyndamax PMS (Other: Alias Study Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: ATTR-CM (Transthyretin Amyloid Cardiomyopathy)
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Adults diagnosed with transthyretin-mediated amyloidosis (ATTR-CM)
  Interventions: Drug: Vyndamax (tafamidis 61mg)

INTERVENTIONS:
Drug: Vyndamax (tafamidis 61mg) — As prescribed in real world practice
  Other Names: Tafamadis

SUMMARY:
This non-interventioal study will be performed by design of post-marketing surveillance (PMS) as an additional pharmacovigilance activity of the Risk Management Plan (RMP) for Vyndamax® Capsules, which is required by the Ministry of Food and Drug Safety (MFDS) according to the local regulation. This post-marketing surveillance will investigate the safety and effectiveness of Vyndamax® Capsules as the treatment of transthyretin amyloid cardiomyopathy during 10 years under the setting of routine practice in Korea.

ELIGIBILITY:
*Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* 1. Adult patients with the cardiomyopathy of wild type or hereditary transthyretin-mediated amyloidosis (ATTR-CM)
* 2. Patients to whom Vyndamax® Capsules is prescribed for the treatment of the cardiomyopathy of wild type or hereditary transthyretin-mediated amyloidosis (ATTR-CM)
* 3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

  * Exclusion criteria

Patients meeting any of the following criteria will not be included in the study according to the local product label:

* 1. Patient with hypersensitivity or case history to tafamidis or to any of the excipients in the product
* 2. This product contains sorbitol (E420). Patients with rare hereditary problems of fructose intolerance should not take this medicine.
* 3. Patient who has a contraindication to Vyndamax® Capsules according to the approved local product label

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in patients who have received at least 1 dose of Vyndamax Capsules for the following indications as per local product label.(Treatment of the cardiomyopathy of wild type or hereditary transthyretin-mediated amyloidosis (ATTR-CM) in adults to reduce cardiovascular mortality and cardiovascular-related hospitalization)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Adverse Events (AEs) | Baseline through 6 months of treatment
  The primary interest of this study is the incidence of AEs investigated during administration period and within 28 days after discontinuation of Vyndamax® Capsules. Incidence of AEs, 95% confidence interval and the number of AEs will be presented.
  Serious AEs/ADRs, unexpected AEs/ADRs, unexpected serious AEs/ADRs will be summarized separately table.

SECONDARY OUTCOMES:
Change from baseline in the New York Heart Association (NYHA) class at Month 6 | Baseline, month 6
Change from baseline in the 6 Minute Walk Distance (6MWD) at Month 6 | Baseline, month 6
Global assessment by investigator at Month 6 | Baseline, month 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461080